CLINICAL TRIAL: NCT07037251
Title: Screening for Fibromyalgia Among Patients With Suspected Endometriosis
Status: Recruiting | Type: Observational
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 0129-23-AAA
Record Dates: First submitted 2024-05-19; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia; Endometriosis
Keywords: fibromialgia; endometriosis
MeSH Terms: conditions — Fibromyalgia; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: there is no intervention — there is no intervention only observation

SUMMARY:
The main purposes of the study are:

To determine the prevalence of fibromyalgia among patients with suspected endometriosis during their initial visit to an endometriosis clinic.

Secondary aims include staging of endometriosis in these patients according to the AAGL (16,17) endometriosis classification and correlate the prevalence of fibromyalgia with ultrasound and surgical findings. Another aim will be to assess the improvement in symptoms in patients diagnosed with both disorders in comparison to patients with either one separately.

All women with suspected endometriosis will be asked to complete the questionnaire before their first visit to the doctor's office.

Study design

* A single center prospective cohort study
* All patients attending to Endometriosis clinic at Assuta Ashdod University Hospital with suspected endometriosis at initial visit and who will consent and able to sign the consent form for participation.
* Fibromyalgia will be defined by the ACR Preliminary Diagnostic Criteria, including Widespread Pain Index, Symptoms severity scale and somatic symptoms.
* The treating physician will blinded to questionnaire results until the end of the visit.
* At the end of the visit the questionnaire will be analyzed by one of the investigators and if fibromyalgia is found, the patient will also be referred for treatment of this disorder along with the endometriosis treatment.
* Questionnaires will be coded with numbers from 1 to 150.

DETAILED DESCRIPTION:
Screening for fibromyalgia among patients with suspected endometriosis Introduction Fibromyalgia is a chronic pain syndrome affecting mainly females. Most patients have soft tissue sensitivity and pain, without any abnormality indicating inflammation or damage to those tissues. Therefore, diagnosis of the disease is made promptly by ruling out other conditions and assessing the patients with physical examination and designated thorough questionnaires. For epidemiological purposes the common questionnaire is the London Fibromyalgia Epidemiology Study Screening Questionnaire (LFESSQ) based on pain and fatigue criteria, without referring to tender points. The most recent and practical questionnaire for diagnosing and assessing the severity of the syndrome is the Modified ACR Preliminary Diagnostic Criteria, first published in 2011 and revised in 2016. A patient that fulfills the diagnostic criteria according to the questionere can be diagnosed with this condition without need for other tests.

The pathophysiology of fibromyalgia is not well understood, however is has been extensitvely studied. It is suggested that changes in central pain modulation cause widespread pain and it is associated withseveral genetic and environmental risk factors. This phenomenon of central sensitization also plays a role in chronic pain in patients with endometriosis.

Fibromyalgia and its relation to endometriosis have been studied. Similarly to fibromyalgia, endometriosis is associated with chronic pain and comorbidities. Greenbaum et al. found that endometriosis and fibromyalgia are both associated with autoimmune diseases, such as inflammatory bowel disease and rheumatic arthritis. In addition, both conditions are known to reduce the quality of life and have been associated with depressive symptoms. A study by Nunes et al examined whether there is a difference in the prevalence of fibromyalgia among healthy women or those diagnosed with endometriosis. They did not find any difference in the prevalence between the two groups, however they did identify that the quality of life among women diagnosed with endometriosis was poorer. Another study by Coloma et al. found that there is a higher prevalence of fibromyalgia among women diagnosed with deep infiltrating endometriosis using the LFESSQ, and once again poorer quality of life. Diagnosing fibromyalgia in patients with endometriosis might impact our treatment in these patients, enabling us to better address their pain and offer more focused treatment.

As far as we know, no study was performed in order to assess the prevalence of fibromyalgia in patients with suspected endometriosis as part of their initial visit.

Objectives:

The main purposes of the study are:

To determine the prevalence of fibromyalgia among patients with suspected endometriosis during their initial visit to an endometriosis clinic.

Secondary aims include staging of endometriosis in these patients according to the AAGL endometriosis classification and correlate the prevalence of fibromyalgia with ultrasound and surgical findings. Another aim will be to assess the improvement in symptoms in patients diagnosed with both disorders in comparison to patients with either one separately.

All women with suspected endometriosis will be asked to complete the questionnaire before their first visit to the doctor's office.

Study design

* A single center prospective cohort study
* All patients attending to Endometriosis clinic at Assuta Ashdod University Hospital with suspected endometriosis at initial visit and who will consent and able to sign the consent form for participation.
* Fibromyalgia will be defined by the ACR Preliminary Diagnostic Criteria, including Widespread Pain Index, Symptoms severity scale and somatic symptoms.
* The treating physician will blinded to questionnaire results until the end of the visit.
* At the end of the visit the questionnaire will be analyzed by one of the investigators and if fibromyalgia is found, the patient will also be referred for treatment of this disorder along with the endometriosis treatment.
* Questionnaires will be coded with numbers from 1 to 150.

Inclusion criteria All women with suspected endometriosis in their first visit to endometriosis clinics in Assuta Ashdod Hospital Exclusion criteria Proven fibromyalgia prior to the first visit. Sample size According to previous studies , have used a sample size of 229 patients ,difference between fibromyalgia prevalence in patients with and without endometriosis 6,7% (CI 1.8 -20.5) we assume that 150 eligible cases will be found sufficient ( with 80% power and 5% significance level) Statistical analysis: results will be summarized in Excel table and then analyzed by statistician and the investigators.

ELIGIBILITY:
Inclusion Criteria:

* All women with suspected endometriosis in their first visit to endometriosis clinics in Assuta Ashdod Hospital

Exclusion Criteria:

* Proven fibromyalgia prior to the first visit.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women
Study Population: All women with suspected endometriosis in their first visit to endometriosis clinics in Assuta Ashdod Hospital
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Fibromyalgia in patients with endometriosis | within 2 years from the beginning of the study
  Occurrence of Fibromyalgia on first visit to endometriosis clinic

SECONDARY OUTCOMES:
staging of endometriosis in these patients according to the AAGL (16,17) endometriosis classification and correlate the prevalence of fibromyalgia with ultrasound and surgical findings. | The questionnaire will be annalized at the end of the study, within 2 years of initial visit
  staging of endometriosis in these patients according to the AAGL (16,17) endometriosis classification and correlate the prevalence of fibromyalgia with ultrasound and surgical findings.
To determine the prevalence of fibromyalgia among patients with suspected endometriosis during their initial visit to an endometriosis clinic. | questionnaire for fibromialgia will be filled up to one day from visit to clinic
  Patients will fill diagnostic questionnaire for fibromialgia that will be analyzed by rheumatologists. To determine the prevalence of fibromyalgia among patients with suspected endometriosis during their initial visit to an endometriosis clinic.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Ashdod University Hospital, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No